CLINICAL TRIAL: NCT03748329
Title: Ultrasound-guided Inferior Alveolar Nerve Block Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Anesthesia Research Foundation (Unknown)
Responsible Party: Principal Investigator, Derek Decloux, Masters Student in Dental Anaesthesiology, University of Toronto
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 34854
Record Dates: First submitted 2017-08-18; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Ultrasound; Local Anesthetic
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Split mouth study
Who Masked: Participant
Masking Description: The transducer will remain in place during the performance of the block but the monitor will be above the head of the patient in the 12 o'clock position so as to not be in direct view.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — Will deposit local anaesthetic intra-orally with the aid of ultrasound to guide the location of the final deposition.

SUMMARY:
The primary objective is to compare the success of the inferior alveolar nerve block using ultrasound versus a traditional landmarking technique (which historically has an approximate failure rate as high as 33.8%). The secondary objective is to demonstrate that delivering a block under ultrasound guidance does not cause any additional pain to patients, as well as to reconfirm data shown in a previous study that the intra-oral transducer is well-tolerated among patients.

DETAILED DESCRIPTION:
Inferior alveolar nerve blocks are necessary to perform dental procedures in the mandible. The standard mandibular block (also known as the Halsted Technique, or the Inferior Alveolar Nerve Block) is based on intraoral landmarks but due to anatomical variation between patients, the failure rate, and therefore incomplete anaesthesia of the mandibular teeth, is high. Success rates have been reported anywhere from 66.2%-96.5% (Montagnese, 1984). Different approaches have been described to improve the success of blocking the inferior alveolar nerve but all have had varying rates of success (Blanton, 2002; Todorovic, 1986). Regardless, none are able to consistently and reliably block the inferior alveolar nerve one-hundred percent of the time.

Ultrasound is a valuable clinical tool to improve the accuracy of nerve blocks, and is also an important teaching tool. Ultrasound imaging is capable of identifying the relevant anatomy in the region of interest and has become common place during placement of spinal nerve blocks and many commonly recognized peripheral nerve blocks (Denny et Harrop-Griffiths, 2005). In studies of peripheral nerve blockade of the spine, the use of ultrasound should be able to reduce the number of needle passes required to achieve anaesthesia of a peripheral nerve and has been shown to reduce procedural times (Griffin et Nicholls, 2010). In addition, onset of sensory blockade is faster because of more intimate proximity of the needle tip to the nerve. Finally, the ability to visualize, and thereby ensure, the spread of local anaesthetic around the nerve also aids in the speed of onset of the block (Griffin et Nicholls, 2010). However, ultrasound has yet to be used successfully in intraoral trigeminal nerve blocks.

While Hannan et al. (1999) did compare ultrasonography to traditional landmarking for the inferior alveolar nerve block, there was no increase in success of the block. It should be noted that Hannan et al. was unable to visualize the nerve and instead used the inferior alveolar artery as a surrogate landmark to approximate proximity to the inferior alveolar nerve. Since the study by Hannan et al., there have been marked improvements to ultrasound hardware, i.e. transducers, and software, i.e. processors, to improve resolution and increase the ability to differentiate objects in soft tissue, specifically the neural structures from the vascular structures.

The inferior alveolar nerve itself can now be visualized by ultrasound in unembalmed human cadavers and can be accurately targeted with a needle by placing dye around the inferior alveolar nerve and confirmed by dissection performed by a blinded anatomist (Chanpong, 2013). The same study had a clinician consistently identify the inferior alveolar nerve bilaterally in 20 living individuals by ultrasound. In addition, according to the satisfaction survey performed, the intraoral ultrasound probe was just as comfortable as a bite block placed on the contralateral side. Based on a 10 point Likert scale (1 being very uncomfortable and 10 being very comfortable), the ultrasound probe scored a mean of 7.3 and the bite block a 7.5, and all 20 volunteers were able to complete bilateral scans. Given that the inferior alveolar nerve block can be easily visualized by ultrasound, the accuracy of needle placement may be significantly improved.

Adjacent to the inferior alveolar nerve are the inferior alveolar artery and the inferior alveolar vein. The risk of inadvertent vascular puncture of these vessels while performing an Inferior Alveolar Nerve Block has been reported to be anywhere from 2.6% to 30% (Malamed, 2013). By being able to guide the needle using ultrasound, the incidence of their puncture, and incidence of nerve puncture, may also be reduced.

Finally, it has been noted that when patients experience a painful "electric shock"-like symptom during mandibular block anaesthesia, these events may be a result from direct contact to the lingual nerve (Harn et Durham, 1990). This sensation is said to occur approximately seven percent of the time during mandibular blocks and can be associated with persistent reduced sensation to the trigeminal nerve. Avoiding direct insult to any of the surrounding nerves would reduce intra-operative pain to the patient during inferior alveolar nerve blockade.

In summary, ultrasound-guided inferior alveolar nerve block is a novel technique that may improve the success of the nerve block and reduce inadvertent puncture of surrounding structures. Currently, there is no published description of the use of ultrasound to guide precise needle placement to adjacent proximity of the inferior alveolar nerve to accomplish blockade of the respective nerve in living patients.

ELIGIBILITY:
Inclusion criteria include male and female volunteers been the ages of 18 and 65 years old who can understand the study protocol and are able to give consent. Subjects must weigh between 40 kg and 100kg and fall under the American Society of Anesthesiology (ASA) classification I or II. At least one unrestored tooth distal to the lateral incisor must be present in both mandibular quadrants for EPT testing. Participants must also be able to open their mouth sufficiently to place a transducer and needle against the medial mandibular ramus.

Exclusion criteria include volunteers with serious medical conditions (ASA 3 or higher). Pregnant volunteers and those who have an allergy to mepivicaine or are on systemic anticoagulation will be excluded. Volunteers with infections, lesions, or anatomic anomalies at the site of the injection or have a pre-existing neurologic deficit in the mouth, head, or neck will also be excluded. Other exclusion criteria include volunteers who have taken any CNS depressants, opioids, non-steroidal anti-inflammatories, and/or acetaminophen in the 48 hours prior to testing. Subjects who are unable to speak English AND are unable to provide their own interpreter at all necessary appointments (screening, data collection, follow-up phone call) will be excluded as the data collection requires direct communication with one of the investigators (they are only English speaking) to discuss consent, instruction in the study, and possible post-operative adverse events and their associated management.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Ultrasound vs Traditionally Landmarked Method | Immediate
  Compare the success of the inferior alveolar nerve block using ultrasound versus a traditional landmarking technique using pulpal anaesthesia as assessed by an electric pulp tester.

SECONDARY OUTCOMES:
Pain | Immediate
  Demonstrate that delivering a block under ultrasound guidance does not cause any additional pain to patients comparing techniques using a 100mm VAS.
Comfort of ultrasound | Immediate
  Reconfirm data shown in a previous study that the intra-oral transducer is well-tolerated among patients comparing techniques using a 100mm VAS.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No